CLINICAL TRIAL: NCT05774119
Title: Effect of Coffee Consumption on Hunger, Satiety, and Appetite-regulating Hormones in Women With Overweight or Obesity
Brief Title: Effect of Coffee Consumption on Appetite Traits in Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Livier Nathaly Torres Castillo, Associate Professor B, University of Guadalajara
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CI-03421
Record Dates: First submitted 2022-11-01; First posted 2023-03-17 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Obesity
Keywords: coffee; hunger; ghrelin; cholecystokinin
MeSH Terms: conditions — Obesity | interventions — Breakfast; Coffee; Water

STUDY DESIGN:
Intervention Model Description: Crossover randomized clinical trial. Premenopausal women with overweight or with obesity will be included. The participants attend 3 sessions: in the first, a clinical history is applied, and anthropometric measurements are taken; in the second and third sessions they consume a standard breakfast (519 kcal) together with 240 ml of coffee with 6 mg/caffeine/kg of weight or the same breakfast but accompanied by 240 ml of water. The sequence of the type of intervention is randomly assign with a period of 1 week wash. Fasting and every 30 minutes during the 3 hours following breakfast consumption, sensations of appetite are recorded using visual analog scales. Fasting, 30 and 180 min after breakfast consumption, ghrelin and cholecystokinin levels are measured. Dietary intake is recorded on the day before the two interventions and on the day of intervention, after breakfast consumption.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- breakfast with coffee (Experimental): 250 mL of water with 6 mg/caffeine/kg
  Interventions: Other: breakfast with coffee
- breakfast with water (Placebo Comparator): 250 mL of water
  Interventions: Other: breakfast with water

INTERVENTIONS:
Other: breakfast with coffee — breakfast with coffee with 6 mg/caffeine/kg body weight
  Arms: breakfast with coffee
Other: breakfast with water — breakfast with 250 mL of water
  Arms: breakfast with water

SUMMARY:
The effect of coffee consumption on appetite is not clear, there are studies that show an effect on the regulation of energy intake, reducing hunger and/or increasing satiety. The purpose of this trial is to evaluate the effect of 6 mg/caffeine/kg of body weight on hunger, satiety, dietary intake, biochemical variables and ghrelin and cholecystokinin concentration in overweight and obese women.

DETAILED DESCRIPTION:
Randomized crossover clinical trial to be realized in women between 20 and 40 years of age with overweight or obesity and apparently healthy who reside in the city of Guadalajara, Jalisco.

Their participation involves their attendance to 3 interventions, in the first one it is verified whether or not they meet the inclusion criteria, a clinical history is applied to take information on pathological history, clinical data, nutritional aspects, sociodemographic and lifestyle aspects and anthropometric measurements; then they are randomly assigned to the two types of interventions in the next two subsequent ones.

In the second and third interventions (with an interval of 7 days between them), participants will attend in the follicular phase of their menstrual cycle during the experiments to avoid variability in appetite.

They will arrive at the institute at 8 am after an overnight fast, consume a standard 400 kcal breakfast with a distribution of 55% carbohydrates, 30% lipids and 15% protein. along with 240 ml of coffee with 6 mg/caffeine/kg body weight or the same breakfast, but with 240 ml of water.

On an empty stomach and every 30 min during the 3 h following the consumption of breakfast with the beverage, the participants recorded their level of hunger, fullness, satiety, desire to eat and prospective consumption, desire to eat specific foods: sweet, salty, fatty, tasty, and sed through visual analog scales (VAS).

On an empty stomach, 30 minutes after consuming breakfast with the beverage and after 180 min, a blood sample will be taken from which serum will be obtained for glucose, total cholesterol, HDL cholesterol, LDL cholesterol, VLDL cholesterol, triglycerides, ghrelin and cholecystokinin determinations.

In the first intervention, participants will be instructed to fill out a 24-hour reminder form to assess dietary intake, and will be asked to record all food and beverages consumed for 3 days prior to the two interventions. Participants will also be instructed to fill out a 24-hour post-breakfast reminder with or without coffee.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20 and 40 years old
* Body mass index between 25-40 kg/m2.
* Regular menstrual cycle of 23-32 days in the last 3 months.
* Moderate consumption of coffee (up to 4 cups per day)
* Having the habit of eating breakfast
* Availability of time in the morning

Exclusion Criteria:

* Use of any type of contraceptives in the last three months.
* Use of hypoglycemic, lipid-lowering, weight-loss, appetite altering and psychiatric medications.
* Diagnosis of diabetes mellitus, hypertension, cancer, polycystic ovary syndrome, hypothyroidism, hyperthyroidism, infectious disease, renal disease, dysgeusia, and gallbladder disease.
* Weight loss ≥5% of their weight in the last 6 months.
* Consumption of more than 20 g of alcohol per day.
* Smoking
* Pregnant or breastfeeding
* vegetarian or vegan

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in ghrelin concentration | Baseline, at 30 minutes postprandially, and at 180 minutes postprandially.
  Ghrelin hormone measured by ELISA assay (Enzyme-Linked ImmunoSorbent Assay) according to the manufacturer's recommendations. The kit is GHRL/Ghrelin ELISA Kit catalog number ELH-GHRL. Ghrelin is measured in pg/mL.
Change in cholecystokinin concentration | Baseline, at 30 minutes postprandially, and at 180 minutes postprandially.
  Cholecystokinin measured by ELISA assay (Enzyme-Linked ImmunoSorbent Assay) according to the manufacturer's recommendations. The kit is Human CCK Enzyme Immunoassay Kit catalog number EIA-CCK-1. Cholecystokinin is measured in pg/mL.
Change in dietary intake | Post intervention, the following 24 hours after finishing the intervention
  Analysis of the 24 hour dietary intake recall consumed the rest of the day after the intervention. Analyzed with the Nutritionist Pro TM Software.
Change in appetite feelings | Baseline and in the following 180 minutes postprandially, measured every 30 minutes.
  Hunger, fullness, satiety, desire to eat and prospective consumption are assessed with the visual analog scales (VAS). They are composed of 100 mm long lines, where at one end the term "None" or "Not at all" is placed and at the other end the term "Yes, a lot" or "As much as I have never felt". The patient marks a point between these two extremes and quantification is done by measuring the distance from the left end of the line to the mark which is scored.
Change in desire for specific types of food | Baseline and in the following 180 minutes postprandially, measured every 30 minutes.
  The desire to eat specific foods: sweet, salty, fatty, tasty and thirsty, was evaluated with visual analog scales, consisting of lines in which at one end is placed the term "Yes, very much" and at the other end the term "No, not at all". The patient marks a point between these two extremes and quantification is done by measuring the distance from the left end of the line to the mark, to which a score is given.

SECONDARY OUTCOMES:
Change in plasma glucose | Baseline, at 30 minutes postprandially, and at 180 minutes postprandially.
  Peripheral blood samples were taken by a venous puncture after 12 h of fasting and at 120 min postprandial, and they were immediately centrifuged at 3500 rpm to obtain serum. The serum was separated and stored at -80 ◦C for later use. The concentration of glucose, was measured with a dry chemistry analyzer "Vitros 350 Chemistry" (Ortho-Clinical Diagnostics, Johnson & Johnson Services Inc., Rochester, NY, USA).
Change in lipid profile: total cholesterol, triglycerides, high density lipoprotein, low-density lipoprotein, very low-density lipoprotein | Baseline, at 30 minutes postprandially, and at 180 minutes postprandially.
  Peripheral blood samples were taken by a venous puncture after 12 h of fasting, 30 min and at 180 min postprandial, and they were immediately centrifuged at 3500 rpm to obtain serum. The serum was separated and stored at -80 ◦C for later use. The concentration of triglycerides, total cholesterol, and high-density lipoprotein cholesterol (HDL-c) cholesterol was measured with a dry chemistry analyzer Vitros 350 Chemistry (Ortho-Clinical Diagnostics, Johnson & Johnson Services Inc., Rochester, NY, USA). Low-density lipoprotein cholesterol (LDL-c) was calculated with the Friedewald formula, except when triglycerides levels were higher than 400 mg/dL. Very-low-density lipoprotein cholesterol (VLDL-c) was calculated as total cholesterol minus the sum of LDL-c + HDL-c.
24 hour dietary intake recall pre-intervention | Baseline
  Analysis of the 24 hour dietary intake recall consumed the day previous to the intervention. Analyzed with the Nutritionist Pro TM Software.
Physical activity | Baseline
  It is evaluated with the International Physical Activity Questionnaire (IPAQ). The questionnaire allows to obtain a quantitative calculation of the MET's (metabolic equivalents), which are a measure that expresses the energetic cost of physical activities. A higher score indicates greater physical activity. The minimum value is 3.3 MET´s /minute/week and there is no a maximum value.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magana-de la Vega L, Martinez-Lopez E, Sanchez-Murguia T, Madrigal-Juarez A, Rodriguez-Reyes SC, Aguilar-Vega I, Torres-Castillo N. Effect of coffee intake on appetite parameters in woman with overweight or obesity: A pilot crossover randomized trial. Endocrinol Diabetes Nutr (Engl Ed). 2024 Jun-Jul;71(6):236-245. doi: 10.1016/j.endien.2024.03.021. PMID 38986627

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT05774119/Prot_SAP_ICF_000.pdf